CLINICAL TRIAL: NCT04306159
Title: Application of Opioid-sparing Multimodal Anesthesia Based on Rectus Sheath Block in Open Upper Abdominal Surgery:A Randomized Controlled Study
Brief Title: Application of Rectus Sheath Block based-on Incision in Upper Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201911
Record Dates: First submitted 2020-02-29; First posted 2020-03-12 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2020-03

CONDITIONS: Opioid Consumption
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General anesthesia (Sham Comparator): Basal blood pressure and heart rate were recorded after midazolam administration of 0.02 mg/kg. Anesthesia was induced with sufentanil 0.4 μg/kg and propofol 2-2.5 mg/kg, IV route. An IV bolus of cisatracurium 0.1 mg/kg IV was given to facilitate tracheal intubation. Anesthesia was maintained with propofol 4-6 mg/kg/h combined dexmedetomidine 0.2 μg/kg/h(after 0.2 μg/kg/h loading dose within 15min)by bispectral index (BIS) 40-60 and additional bolus doses of remifentanil 0.2-0.5 μg/kg/min to keep arterial pressure values around 20% below baseline values. Sufentanil 0.1-0.2 μg/kg and flurbiprofen 100mg was administrated once the abdomen was closed, then a patient controlled analgesia pump was used. No RSB was performed.
  Interventions: Other: General anesthesia
- Subcostal TAP combined with General anesthesia (Experimental): After induction, TAP was performed. The transversus abdominis plane is imaged with the ultrasound probe obliquely on the upper abdominal wall, along the subcostal margin near the midline.The needle tip was advanced to the desired position where 20 mL 0.375%ropivacaine(Dexamethasone 5mg was added)were injected.The technique is repeated on the opposite side. Anesthesia method and management was same as general anesthesia group.
  Interventions: Procedure: Subcostal TAP
- Modified RSB combined with General anesthesia (Experimental): After induction, Modified RSB was performed based on midline incision-guided. The rectus muscle is imaged with the ultrasound probe in a transverse orientation below the xiphisternum and above the umbilicus.The needle tip was advanced to the two desired position where 10 mL ropivacaine 0.375% were injected causing hydrodissection of the rectus muscle away from the posterior rectus sheath.The technique is repeated on the opposite side.Anesthesia method and management was same as general anesthesia group.
  Interventions: Procedure: Modified RSB

INTERVENTIONS:
Procedure: Subcostal TAP — Subcostal transversus abdominis plane block
  Arms: Subcostal TAP combined with General anesthesia
Procedure: Modified RSB — Rectus Sheath Block under the guidance of surgical incision
  Arms: Modified RSB combined with General anesthesia
Other: General anesthesia — Traditional general anesthesia management
  Arms: General anesthesia

SUMMARY:
General anesthesia combined subcostal transversus abdominis plane (TAP)or rectus sheath block (RSB)can significantly reduce the use of opiates in minimally invasive surgery.However, similar reduction was not observed in open abdominal surgery during perioperative period.Therefore, the investigators should try to improve the blocking methods to reduce the side effects of a large number of opiates. Based on the range and its analgesic effect of various nerve block is obviously related to the injection site of local anesthetics, this randomized controlled study hypothesized that modified RSB under the guidance of surgical incision may be more effective in inhibiting the harmful stimulation of surgery.

DETAILED DESCRIPTION:
For abdominal cancer surgery with midline incision, subcostal transversus abdominis plane or rectus sheath block combined with general anesthesia was more effective in reducing pain scores and opioid consumption compared with general anesthesia alone. However, there was no statistically significant difference in supplementary fentanyl during operation. Besides adequate pain relief around incisions, blunting visceral traction response has also an important role in hemodynamic stability.With the evidences for a potential mechanism for the antinociceptive effects of propofol on visceral nociception and dexmedetomidine combined with oxycodone can provide good visceral analgesia, the investigators supposed that visceral nociception was well suppressed by adequate antinociceptive drugs. The propofol combination with dexmedetomidine may had significant effect on the reduction of the sympathoadrenergic tone with decrease of blood pressure and heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85 years
* Anesthesiologists (ASA) risk classification I to IV
* Scheduled to undergo midline incision of upper abdomen (From xiphoid to navel )

Exclusion Criteria:

* Patient refusal
* Any contraindications to regional techniques (allergy to local anesthetics, infection around the site of the block, and coagulation disorder)
* History of analgesics dependence
* Any difficulty with communication
* Allergy to the study drugs
* Heat rate < 50 beats/minutes or II-III Atrioventricular block
* Previous open surgery
* Previous definite history of malignant tumor
* Who had an estimated intraoperative blood loss of more than 500 mL

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Opiate consumption | From the beginning to the end of anesthesia,up to 6 hours.
  Remifentanil consumption
Tumor recurrence rate | 1-year after surgery
  Tumor recurrence rate after surgery

SECONDARY OUTCOMES:
Opiate consumption | From the end of anesthesia to 48 hours after surgery, up to 2 days.
  Sufentanil consumption
Pain scores | 2 hours after surgery
  1. Through visual analogue scale (from 0 to 10) to assess the degree of pain;
  2. The number 0 means no pain and the number 10 means the most pain;
  3. Patients with visual analogue scale greater than 3 points should have remedial analgesic drugs.
Pain scores | 6 hours after surgery
  1. Through visual analogue scale (from 0 to 10) to assess the degree of pain;
  2. The number 0 means no pain and the number 10 means the most pain;
  3. Patients with visual analogue scale greater than 3 points should have remedial analgesic drugs.
Pain scores | 12 hours after surgery
  1. Through visual analogue scale (from 0 to 10) to assess the degree of pain;
  2. The number 0 means no pain and the number 10 means the most pain;
  3. Patients with visual analogue scale greater than 3 points should have remedial analgesic drugs.
Pain scores | 24 hours after surgery
  1. Through visual analogue scale (from 0 to 10) to assess the degree of pain;
  2. The number 0 means no pain and the number 10 means the most pain;
  3. Patients with visual analogue scale greater than 3 points should have remedial analgesic drugs.
Pain scores | 36 hours after surgery
  1. Through visual analogue scale (from 0 to 10) to assess the degree of pain;
  2. The number 0 means no pain and the number 10 means the most pain;
  3. Patients with visual analogue scale greater than 3 points should have remedial analgesic drugs.
Pain scores | 48 hours after surgery
  1. Through visual analogue scale (from 0 to 10) to assess the degree of pain;
  2. The number 0 means no pain and the number 10 means the most pain;
  3. Patients with visual analogue scale greater than 3 points should have remedial analgesic drugs.
Time for first to press pump | Up to 2 days after surgery
  Time for first to press pump
Time of anal exsufflation | Up to 7 days after surgery
  Time for first anal exsufflation
Delirium | Up to 7 days after surgery
  Incidence of postoperative delirium
The occurrence of nausea and vomiting | Up to 7 days after surgery
  Incidence of nausea and vomiting
The occurrence of cardiovascular or cerebrovascular events | From the end of surgery to the time the patients discharge, up to 1 month.
  Incidence of cardiovascular or cerebrovascular adverse events
Length of hospital stay | From the end of surgery to the time the patients discharge, up to 1 month.
  Length of hospital stay
Mortality | 30-day after surgery
  Mortality after surgery
Mortality | 1-year after surgery
  Mortality after surgery
Concentration of norepinephrine | Time before anesthesia induction,immediately after incision,celiac exploration and immediately after closing the abdominal cavity.
  Concentration of norepinephrine during surgery
Concentration of epinephrine | Time before anesthesia induction,immediately after incision,celiac exploration and immediately after closing the abdominal cavity.
  Concentration of epinephrine during surgery
Concentration of cortisol | Time before anesthesia induction,immediately after incision,celiac exploration and immediately after closing the abdominal cavity.
  Concentration of cortisol during surgery
Concentration of tumor necrosis factor-α | Time before anesthesia induction,immediately after incision,celiac exploration and immediately after closing the abdominal cavity.
  Concentration of tumor necrosis factor-α during surgery
Concentration of interleukin-6 | Time before anesthesia induction,immediately after incision,celiac exploration and immediately after closing the abdominal cavity.
  Concentration of interleukin-6 during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guanghong Xu, MD.PHD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China